CLINICAL TRIAL: NCT05978674
Title: The Effect of Rocking Bed on Comfort, Physiological Parameters and Cerebral Oxygenation Level of Preterm Infants: a Near Infrared Spectroscopy Study
Brief Title: The Effect of Rocking Bed on Preterm Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Faculty of Nursing, Selcuk University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukUnı42Konya
Record Dates: First submitted 2023-07-20; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Preterm; Preterm Birth; Nurse's Role
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The study was planned to be conducted in a randomized controlled crossover design. Infants meeting the inclusion criteria will be divided into two groups, group A and group B, according to block randomization. Groups were determined by drawing lots. (A= Rocking bed; B= Jeans) Accordingly, babies included in group A will be taken to the rocking bed first. Babies included in group B will be quoted first. Babies will be laid in these beds for an average of 2 hours. In cross-over design, a washout is recommended in order to control the carry over effect that may result from the interference. We assumed that the total time without interference would be sufficient to control the carryover effect, since the oscillation interference was only applied for half an hour in a two-hour sleep cycle, and there was routine maintenance and feeding cycles between measurements (average 20 min).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: rocking bed group (Experimental): Preterms in the intervention group will lie in a rocking bed for a consecutive two-hour period without treatment and invasive procedures. During 30 minutes of this period, the rocking bed will be in the rocking mode and will stop at the end of 30 minutes.
  Interventions: Behavioral: rocking bed group
- Control Group (No Intervention): Newborns in the control group will be followed in a fixed bed (open bed or incubator).

INTERVENTIONS:
Behavioral: rocking bed group — Babies assigned to the intervention group first will be placed on a rocking bed after routine care such as feeding and diaper changes and when the newborn is stable. A rocking attempt will be applied to the baby placed in the rocking bed for 30 minutes. After 30 minutes, the baby will not be lifted from the bed and will lie in bed for 90 minutes. After a period of two hours in total, the babies will be cared for and fed. Then, babies will be quota and control group measurements will be made.
  Arms: Experimental Group: rocking bed group

SUMMARY:
The study was planned to determine the effect of rocking bed applied to preterm newborns on comfort, physiological parameters and cerebral oxygenase level (rSO2).

DETAILED DESCRIPTION:
In most cultures, providing a newborn baby on the lap or in a rocking bed is mostly used to calm the baby. However, preterm babies who leave the uterus, which is their accustomed environment, in the early period, are positioned on a fixed bed such as an incubator or jeans in the NICU. These beds may reduce the infant's vestibular knowledge and the NICU environment may deprive infants of sensory stimuli. It has been suggested that because the vestibular system is one of the first systems to become functional, preterm infants may be more sensitive to stimulation of the vestibular system than other systems. When the studies were examined, it was seen that limited studies were conducted in the sample of preterm infants and the studies were not recent. Considering that babies are rocked in most cultures, it is thought that the evidence for the effects of the intervention on the baby is insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Born at 32-37 weeks of postmenstruel age
* Not receiving mechanical ventilation support,
* Not receiving analgesia or sedative drug therapy,
* Congenital anomaly, intraventricular hemorrhage, meningitis, chromosomal anomalies, cyanotic congenital heart diseases, neonatal seizures and preterm infants without a diagnosis of sepsis

Exclusion Criteria:

• Infants with diseases that may decrease cerebral oxygenation such as cerebral edema, intraventricular hemorrhage, cerebral hypoxia will be excluded from the study.

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Information Form | First measurement- At 15 minutes after admission in the study
  In the form prepared by the researchers in line with the literature in order to collect introductory information about the baby; There are questions for the baby such as gender, mode of delivery, weight at birth, Apgar score (1st and 5th value), gestational age at birth, postnatal age, weight in the study, diet, type of food, frequency of vomiting (O'Reilly et al., 2011; Provasi et al., 2021; Zimmerman & Barlow, 2012). For the final version of the form, opinions were received from 2 nurses and 1 neonatology specialist, who are experts in pediatric nursing.
COMFORT Scale | First measurement: T0: just before the intervention
  The COMFORT Scale was developed by Ambuel et al. (1992) to determine the comfort and distress of patients in the pediatric intensive care unit. The comfort of the newborn is evaluated through 7 parameters, including muscle tone, calmness/agitation, facial tension, body movements, crying, and respiratory response with YKDS. If the newborn receives mechanical ventilator support, "respiratory response" is scored, and if the newborn is breathing spontaneously, "crying" items are scored. For this reason, the overall scoring of the scale is based on 6 items, and the scores that can be obtained from the scale vary between 6 and 30. A low score from the scale indicates comfort, while an increase in score indicates pain or distress in the newborn (Kahraman et al., 2014; Van Dijk et al., 2009). The Turkish validity and reliability study of YKDS was conducted by Kahraman et al. in 2014 (Kahraman, Başbakal, & Yalaz, 2014).
Newborn Follow-up Form | First measurement: T0: just before the intervention
  This form, created by the researchers, contains information on physiological parameters (heart rate, respiratory rate, and oxygen saturation) and cerebral rSO2 values (Provasi et al., 2021; Zimmerman & Barlow, 2012). The information in the Follow-up Form was evaluated just before the intervention (TO), at the 15th minute of the intervention (T1), at the 30th minute of the intervention (T2), and 15 minutes after the intervention (T3). The form was finalized by taking the opinions of 2 nurses and 1 neonatology specialist, who are experts in pediatric nursing. Physiological parameters of the newborn were followed from the Philips IntelliVue MP40 branded neonatal monitor suitable for neonatal use, and cerebral rSO2 was monitored with the INVOS™ 5100C Cerebral/Somatic Oximeter brand NIRS device available in the clinic.

SECONDARY OUTCOMES:
COMFORT Scale | Second measurement: T1: 15th minute of the intervention
  The COMFORT Scale was developed by Ambuel et al. (1992) to determine the comfort and distress of patients in the pediatric intensive care unit. The comfort of the newborn is evaluated through 7 parameters, including muscle tone, calmness/agitation, facial tension, body movements, crying, and respiratory response with YKDS. If the newborn receives mechanical ventilator support, "respiratory response" is scored, and if the newborn is breathing spontaneously, "crying" items are scored. For this reason, the overall scoring of the scale is based on 6 items, and the scores that can be obtained from the scale vary between 6 and 30. A low score from the scale indicates comfort, while an increase in score indicates pain or distress in the newborn (Kahraman et al., 2014; Van Dijk et al., 2009). The Turkish validity and reliability study of YKDS was conducted by Kahraman et al. in 2014 (Kahraman, Başbakal, & Yalaz, 2014).
Newborn Follow-up Form | Second measurement: T1: 15th minute of the intervention
  This form, created by the researchers, contains information on physiological parameters (heart rate, respiratory rate, and oxygen saturation) and cerebral rSO2 values (Provasi et al., 2021; Zimmerman & Barlow, 2012). The information in the Follow-up Form was evaluated just before the intervention (TO), at the 15th minute of the intervention (T1), at the 30th minute of the intervention (T2), and 15 minutes after the intervention (T3). The form was finalized by taking the opinions of 2 nurses and 1 neonatology specialist, who are experts in pediatric nursing. Physiological parameters of the newborn were followed from the Philips IntelliVue MP40 branded neonatal monitor suitable for neonatal use, and cerebral rSO2 was monitored with the INVOS™ 5100C Cerebral/Somatic Oximeter brand NIRS device available in the clinic.
COMFORT Scale | Third measurement: T2: 30th minute of the intervention
  The COMFORT Scale was developed by Ambuel et al. (1992) to determine the comfort and distress of patients in the pediatric intensive care unit. The comfort of the newborn is evaluated through 7 parameters, including muscle tone, calmness/agitation, facial tension, body movements, crying, and respiratory response with YKDS. If the newborn receives mechanical ventilator support, "respiratory response" is scored, and if the newborn is breathing spontaneously, "crying" items are scored. For this reason, the overall scoring of the scale is based on 6 items, and the scores that can be obtained from the scale vary between 6 and 30. A low score from the scale indicates comfort, while an increase in score indicates pain or distress in the newborn (Kahraman et al., 2014; Van Dijk et al., 2009). The Turkish validity and reliability study of YKDS was conducted by Kahraman et al. in 2014 (Kahraman, Başbakal, & Yalaz, 2014).
Newborn Follow-up Form | Third measurement: T2: 30th minute of the intervention
  This form, created by the researchers, contains information on physiological parameters (heart rate, respiratory rate, and oxygen saturation) and cerebral rSO2 values (Provasi et al., 2021; Zimmerman & Barlow, 2012). The information in the Follow-up Form was evaluated just before the intervention (TO), at the 15th minute of the intervention (T1), at the 30th minute of the intervention (T2), and 15 minutes after the intervention (T3). The form was finalized by taking the opinions of 2 nurses and 1 neonatology specialist, who are experts in pediatric nursing. Physiological parameters of the newborn were followed from the Philips IntelliVue MP40 branded neonatal monitor suitable for neonatal use, and cerebral rSO2 was monitored with the INVOS™ 5100C Cerebral/Somatic Oximeter brand NIRS device available in the clinic.
COMFORT Scale | Fourth measurement: T3: 15 minutes after the end of the intervention
  The COMFORT Scale was developed by Ambuel et al. (1992) to determine the comfort and distress of patients in the pediatric intensive care unit. The comfort of the newborn is evaluated through 7 parameters, including muscle tone, calmness/agitation, facial tension, body movements, crying, and respiratory response with YKDS. If the newborn receives mechanical ventilator support, "respiratory response" is scored, and if the newborn is breathing spontaneously, "crying" items are scored. For this reason, the overall scoring of the scale is based on 6 items, and the scores that can be obtained from the scale vary between 6 and 30. A low score from the scale indicates comfort, while an increase in score indicates pain or distress in the newborn (Kahraman et al., 2014; Van Dijk et al., 2009). The Turkish validity and reliability study of YKDS was conducted by Kahraman et al. in 2014 (Kahraman, Başbakal, & Yalaz, 2014).
Newborn Follow-up Form | Fourth measurement: T3: 15 minutes after the end of the intervention
  This form, created by the researchers, contains information on physiological parameters (heart rate, respiratory rate, and oxygen saturation) and cerebral rSO2 values (Provasi et al., 2021; Zimmerman & Barlow, 2012). The information in the Follow-up Form was evaluated just before the intervention (TO), at the 15th minute of the intervention (T1), at the 30th minute of the intervention (T2), and 15 minutes after the intervention (T3). The form was finalized by taking the opinions of 2 nurses and 1 neonatology specialist, who are experts in pediatric nursing. Physiological parameters of the newborn were followed from the Philips IntelliVue MP40 branded neonatal monitor suitable for neonatal use, and cerebral rSO2 was monitored with the INVOS™ 5100C Cerebral/Somatic Oximeter brand NIRS device available in the clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Küçükoğlu, Prof, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambuel B, Hamlett KW, Marx CM, Blumer JL. Assessing distress in pediatric intensive care environments: the COMFORT scale. J Pediatr Psychol. 1992 Feb;17(1):95-109. doi: 10.1093/jpepsy/17.1.95. PMID 1545324
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] O'Reilly R, Grindle C, Zwicky EF, Morlet T. Development of the vestibular system and balance function: differential diagnosis in the pediatric population. Otolaryngol Clin North Am. 2011 Apr;44(2):251-71, vii. doi: 10.1016/j.otc.2011.01.001. PMID 21474003
- [Background] Provasi J, Blanc L, Carchon I. The Importance of Rhythmic Stimulation for Preterm Infants in the NICU. Children (Basel). 2021 Jul 29;8(8):660. doi: 10.3390/children8080660. PMID 34438551
- [Background] van Dijk M, Roofthooft DW, Anand KJ, Guldemond F, de Graaf J, Simons S, de Jager Y, van Goudoever JB, Tibboel D. Taking up the challenge of measuring prolonged pain in (premature) neonates: the COMFORTneo scale seems promising. Clin J Pain. 2009 Sep;25(7):607-16. doi: 10.1097/AJP.0b013e3181a5b52a. PMID 19692803
- [Background] Zimmerman E, Barlow SM. The effects of vestibular stimulation rate and magnitude of acceleration on central pattern generation for chest wall kinematics in preterm infants. J Perinatol. 2012 Aug;32(8):614-20. doi: 10.1038/jp.2011.177. Epub 2011 Dec 8. PMID 22157627